CLINICAL TRIAL: NCT02990273
Title: The Utility of Thromboelastography in Cirrhotic Patients Undergoing Endoscopic Procedures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding source available which was required for IRB approval
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00113092
Record Dates: First submitted 2016-10-14; First posted 2016-12-13 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Cirrhosis, Coagulopathy
MeSH Terms: conditions — Fibrosis; Hemostatic Disorders | interventions — Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEG (Active Comparator): Blood transfusion
  Interventions: Biological: Blood transfusion
- Prothrombin Time (PT)/International normalized ratio (INR) (Active Comparator): Blood transfusion
  Interventions: Biological: Blood transfusion

INTERVENTIONS:
Biological: Blood transfusion

SUMMARY:
Cirrhosis results in decreased synthesis of both procoagulants and anticoagulants resulting in "rebalanced homeostasis". However, conventional blood tests (platelets/ INR levels) that are performed prior to invasive procedures do not accurately reflect the coagulation changes that occur in cirrhotics, resulting in unnecessary transfusion of blood products. Thromboelastography (TEG) is a global hemostasis assessment tool that is being used in surgery (including liver transplant) to help guide blood product transfusion in the operating room. The investigators would like to compare the use of TEG vs. INR/platelets to help guide blood product transfusion in cirrhotic patients undergoing inpatient endoscopy. The investigators will evaluate to see if there is a decrease in prophylactic blood transfusions prior to endoscopy when using TEG.

ELIGIBILITY:
Inclusion Criteria:

* All 18 yo + cirrhotic patients who are being scheduled for inpatient endoscopy

Exclusion Criteria:

* Patients on blood thinners (prophylactic anticoagulation is permissible)
* Hemodynamically unstable patients requiring pressors (ie ICU level patients)
* Pregnant or lactating individuals
* Inability to provide consent for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

PRIMARY OUTCOMES:
Units of fresh frozen plasma (FFP) and platelet transfused | 2 week
  Will compare how much FFP and platelet transfusion patients receiving between 2 groups.

CONTACTS AND LOCATIONS:
Overall Officials: Tinsay Woreta, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: Undecided